CLINICAL TRIAL: NCT07229001
Title: A Randomized Clinical Trial of Treating Meibomian Gland Disease in a Pediatric Population
Brief Title: Treating Meibomian Gland Disease in a Pediatric Population
Acronym: LLLT in Peds
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Illinois College of Optometry (Other)
Responsible Party: Principal Investigator, Yi Pang, professor, Illinois College of Optometry
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22023
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Dry Eye Disease, Meibomian Gland Disease
Keywords: Dry eye disease, Meibomian Gland Disease
MeSH Terms: conditions — Dry Eye Syndromes; Meibomian Gland Dysfunction | interventions — Lubricant Eye Drops

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- warm compress and artificial tear (Placebo Comparator): warm compress and artificial tear
  Interventions: Other: warm compress and artificial tear
- LLLT (Experimental): LLLT+ warm compress and artificial tear
  Interventions: Other: Low level light treatment

INTERVENTIONS:
Other: Low level light treatment — , LLLT has been confirmed to produced significant improvements in meibomian gland function and symptoms. However, it has not been tested in children. Thus, the study purpose is to determine the treatment effect of LLLT on MGD and DED comparing to using warm compress and artificial tear only in children.
  Arms: LLLT
Other: warm compress and artificial tear — Artificial tears and warm compress have been the traditional treatments for DED.
  Arms: warm compress and artificial tear

SUMMARY:
Dry Eye Disease (DED) is commonly encountered among eye care professionals. DED is a disease of the tears and ocular surface that is multi-factorial resulting in a wide range of symptoms and signs with potentially damaging effects. As technology continues to evolve and as digital devices become more available in social, work environments, and in school settings, patients are increasingly complaining of ocular discomfort and fluctuations in their vision.

In order to diagnose DED which encompasses Meibomian gland dysfunction (MGD), a detailed case history of \patients' symptoms along with imaging to investigate the amount of disease present in their eyes is needed. A customized questionnaire and the Keratograph meibographer will allow for a subjective and objective investigation of dry eye disease in patients. Artificial tears and warm compress are traditional methods used to treat DED. However, many patients continue to have progression of disease. The Marco Equinox Low Level Light Therapy (LLLT) utilizes a LED mask to apply red light to the periorbital and cheekbone regions of the face, which effectively normalizes meibomian gland function. This is a non-invasive treatment of both the upper and lower eyelids, which does not require a gel application. Treatment of both eyes takes approximately 15 minutes. In the clinical studies that have been published, lipid layer interference pattern, non-invasive tear break up time, lissamine green conjunctival staining, Schirmer's test, and upper meibography scores showed significant improvement by 4 weeks after the start of treatment with LLLT. To our knowledge, this has not been studied in the pediatric population, but the disease process is the same. Thus, the study purpose is to determine the treatment effect of LLLT on MGD and DED comparing to traditional treatment (warm compress and artificial tear) only in children.

DETAILED DESCRIPTION:
The clinical diagnosis of Dry Eye Disease is often made using a combination of subjective symptoms and clinical signs. During early development of DED, patients may be asymptomatic. If asymptomatic, the diagnosis of DED is only detectable by the presence of clinical signs. Advanced DED can be debilitating as it can lead to multiple complications including increasing the risk of eye infections and destruction of ocular tissue which eventually causes a loss of functional visual acuity1-3.

Symptoms of dry eye may include ocular itching, burning, redness, irritation, soreness and or edema of the eyelids, foreign body sensation, tearing, fluctuating vision, and contact lens intolerance. The signs of ocular surface damage includes staining to the bulbar conjunctiva and cornea, reduced tear-break-up-time, decreased tear production, and decreased tear quaaulity. Several questionnaires have been reviewed5-6 to assess symptoms of ocular surface disease and dry eye. The Ocular Surface Disease Index (OSDI)5 assesses vision-related function, ocular symptoms, and environmental triggers resulting from dry eye where the goal of the Dry Eye Questionnaire 5 (DEQ-5) is to identify patients with keratoconjunctivitis sicca from those without the condition by asking about the frequency of the feeling of eye dryness. This may be more appropriate to use in the pediatric population as they may not be able to identify with the feeling of dryness, but they should be able to understand 'discomfort' or 'uncomfortable'. While not validated in the pediatric population and regardless of their diagnostic sensitivity for dry eye, standardized questionnaires help assess subjective changes of the patient's symptoms in response to treatment.

Meibomian gland dysfunction can result from a variety of factors, including but not limited to incomplete blinking due to the gland not being able to express a clear lipid layer. This can result in inadequate distribution of the lipid component of the tear layer thereby disrupting adherence of the tears to the eye and thus causing patients to experience the common symptom of "dry eyes." 1,3,4 Once atrophy of the gland occurs, the damage cannot be reversed. Therefore, it is crucial for these patients to maintain healthy tear films and meibomian glands so they don't experience a decrease in visual acuity that can interfere with activities of daily life.

There are several factors which have been proposed to decrease the quality the tear layer and affect the viability of the meibomian glands, and they will be assessed during this study via questionnaires. The one of main interest, particularly in the pediatric population is digital device use. Patient usage of digital devices including: handheld tablets, smart phones, laptops, and computers are increasing as new technology develops and as social and work environments adapt to these technological changes. With the increase in usage of digital devices, eye care practitioners have noted an increase in dry eye signs and symptoms. The potential adverse effect of increased digital device usage may interfere with work performance, productivity, and quality of life.7-9

High levels of mild meibomian gland atrophy have been reported in the pediatric population. This may be due to increased digital device use and near demands of schoolwork. Subsequently, we should be examining young patients for meibomian gland atrophy and dysfunction as early as possible as it may have implications for future development of dry eye disease and complications. Artificial tears and warm compress have been the traditional treatments for DED. Recently, LLLT has been confirmed to produced significant improvements in meibomian gland function and symptoms.10 However, it has not been tested in children. Thus, the study purpose is to determine the treatment effect of LLLT on MGD and DED comparing to using warm compress and artificial tear only in children.

ELIGIBILITY:
Inclusion Criteria:

* subjects with severe MGD

Exclusion Criteria:

* i. Thyroid disease ii. Autoimmune disease iii. Diabetes iv. History of ocular surgery other than refractive surgery v. Disfiguring eye trauma vi. Active infections or severe allergic conjunctivitis vii. Currently pregnant or nursing viii. Epilepsy vii.ix. Migraine

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in MG | 1 months
  atrophy score
MG score | 1 month
  atropine score

CONTACTS AND LOCATIONS:
Locations (1):
- Illinois College of Optometry, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided